CLINICAL TRIAL: NCT02853162
Title: Ablative tReatment of Inoperable REnal Cell Carcinoma Using STereotactic Body Radiotherapy (ARREST-study)
Acronym: ARREST
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, L.G.W. Kerkmeijer, MD, PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL55770.041.15
Record Dates: First submitted 2016-06-24; First posted 2016-08-02 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Stereotactic body radiotherapy; MRI; Renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARREST-study (Experimental): SBRT renal cell carcinoma 5 times 7Gy
  Interventions: Radiation: ARREST-study

INTERVENTIONS:
Radiation: ARREST-study — Radiotherapy will be delivered in five fractions of 7 Gy every other day. An additional contrast enhanced MRI scan will be performed after the 2nd treatment fraction, and after 6 and 12 months

SUMMARY:
Phase II study (n=30) to evaluate the safety and feasibility of stereotactic body radiation therapy (SBRT) with fiducial markers in inoperable patients with renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
Rationale: The standard treatment of RCC is (partial-) nephrectomy. Alternatives to this treatment are less invasive techniques like radio frequency ablation (RFA) and cryoablation (CA). Stereotactic body radiation therapy (SBRT) is an alternative curative treatment modality, which has shown promising results in several North-American phase I-II studies over the last years. In this study, we aim to evaluate the safety and feasibility of SBRT for patients with inoperable RCC on a conventional cone beam computed tomography (CBCT) linear accelerator.

Objective: To evaluate safety and feasibility of stereotactic body radiation therapy (SBRT) with fiducial markers in inoperable patients with renal cell carcinoma (RCC).

Study design: Single arm prospective study. Study population: Inoperable patients ≥ 18 years, with a pathology proven RCC fulfilling the inclusion criteria.

Intervention: Prior to treatment, patients will undergo fiducial marker placement (in combination with a biopsy, if RCC has not been pathology proven), followed by a contrast enhanced planning computed tomography (CT)-scan and a contrast enhanced MRI-scan. Fiducial markers will be used as this increases visibility of the tumor and therefore the accuracy of radiotherapy, particularly the irradiated healthy kidney tissue will be diminished by using this approach. Baseline toxicity and quality of life will be assessed.

SBRT using a VMAT technique will be delivered in five fractions of 7 Gy every other day. The target volume for treatment is defined on a 4D planningCT and MRI and the tumor is treated in the midposition of the breathing cycle. After treatment, follow-up will be at 1, 3, 6 and 12 months at the Radiotherapy department, followed by standard follow-up by the urologist. An additional contrast enhanced MRI scan will be performed after the 2nd treatment fraction, and after 6 and 12 months to assess treatment response to prepare for future MR-guided (MR-linac) radiotherapy. Toxicity and quality of life will be assessed during follow-up.

Main study parameters/endpoints: Newly developed acute toxicity grade 3 or more according to the Common Terminology Criteria for Adverse Events (CTC-AE) version 4.0.

The treatment is considered successful if all 5 treatments are completed and if in total <15% of the patients (=5 patients) report a toxicity ≤ grade 3.

Secondary endpoints will be treatment response, (late) toxicity assessment, local control rate and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Inoperability, or when a patient refuses surgery (i.e. not eligible for (partial-) nephrectomy or RFA);
* Kidney function allows for intervention, as evaluated by treating urologist (taking into account eGFR and renogram);
* Age ≥ 18 years;
* Written informed consent;
* Diagnosis of RCC confirmed by pathology (in case determined after informed consent, patients who are not eligible anymore (no RCC) will be excluded).

Exclusion Criteria:

* Evidence of metastatic disease;
* Exclusion criteria for contrast enhanced MRI scan, according to the protocol of the department of Radiology, UMC Utrecht;
* Patients with one functioning kidney;
* Prior renal surgery (partial nephrectomy);
* Prior radiotherapy on upper abdomen;
* Unsafe to have fiducial marker implantation: i.e. anticoagulant agents use other than acetylsalicyl acid, which cannot be safely stopped/bridged for implantation:
* WHO ≥ 3.
* Chemotherapy < 3 weeks before treatment;
* Targeted therapy (sunitinib, etc.) ≤ 7 days before treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events grade >2 as assessed by CTCAE v.4.0 | Within 90 days after radiotherapy
  The treatment is considered successful if all 5 treatments are completed and if in total <15% of the patients (=5 patients) report an acute toxicity ≤ grade 3

SECONDARY OUTCOMES:
Radiological response | 5 years after radiotherapy
  Radiological treatment response of the tumor, measured according to the RECIST criteria, in combination with functional imaging parameters (multiparametric MRI).
Number of participants with correlation of functional MRI (DCE and DWI) changes during treatment and radiological response after treatment | 12 months after radiotherapy
  Response prediction (contrast enhanced MRI during treatment, after 2nd fraction)
Disease specific survival | 5 years after radiotherapy
  Disease specific survival
Acute and late toxicity | 5 years after radiotherapy
  Common Terminology Criteria for Adverse Events (CTC-AE) version 4.0
Quality of life questionnaire | 12 months after radiotherapy
  EORTC-QLQ-C30
Overall survival | 5 years after radiotherapy
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: L GW Kerkmeijer, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided